CLINICAL TRIAL: NCT07126769
Title: Virtual Knowledge, Real Stress: The Role of Cyberchondria Severity in Women Undergoing Infertility Treatment
Brief Title: Cyberchondria and Stress in Women Undergoing Infertility Treatment
Status: Recruiting | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Güzin Ünlü Suvari, Lecturer, Acibadem University
Other Study IDs: 2025-07/272
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Cyberchondria; Stress; Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study examines how searching for health information on the internet may affect stress and emotional well-being in women undergoing infertility treatment. Infertility is a common condition that impacts about 48 million couples worldwide and can cause not only physical challenges but also significant emotional strain, including anxiety, depression, and stress. Many women turn to the internet to seek answers about their condition and treatment. While online information can be helpful, it is not always accurate or consistent, which can increase worry and confusion. This repeated and sometimes excessive searching for health information, known as "cyberchondria," has been linked in previous research to increased stress and anxiety. This study will assess women's online information-seeking patterns, infertility-related stress, and overall emotional and social well-being, aiming to better understand the role of cyberchondria in the infertility treatment process. The results may help healthcare professionals offer more targeted support and guidance to women facing these challenges.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing infertility treatment and those who have experienced various treatment methods (IUI, IVF, ICSI).
* Women willing to participate in the study.
* Women who understand and speak Turkish.

Exclusion Criteria:

* Women with psychological disorders (e.g., clinical depression, anxiety disorders).
* Women not undergoing infertility treatment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women aged 18 to 45 undergoing infertility treatment (IUI, IVF, ICSI), who speak Turkish, consent to participate, and have no psychological disorders.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | At baseline (one-time assessment at enrollment)
  This form includes 24 questions divided into four sections covering women's sociodemographic details, health information, digital health search behaviors, and reproductive health.
Screening Tool on Distress in Fertility Treatment (SCREEN-IVF) | At baseline (one-time assessment at enrollment)
  A 28-item scale assessing psychosocial risk factors in individuals undergoing infertility treatment. It includes subscales for anxiety, social support, helplessness, acceptance, and depression. Scores above specific cutoff points indicate elevated risk levels in these areas.
Infertility Stress Scale | At baseline (one-time assessment at enrollment)
  Consists of 14 items across three subscales: Personal Stress (6 items), Marital Stress (4 items), and Social Stress (4 items). Higher scores reflect increased stress levels. Items are rated on Likert scales, with score ranges for each subscale indicating the severity of stress.
Short Form of the Cyberchondria Severity Scale | At baseline (one-time assessment at enrollment)
  A 12-item scale measuring severity of excessive online health searches, covering Excessiveness, Distress, Reassurance, and Compulsion subscales. Items scored on a 5-point Likert scale. Higher total scores indicate greater cyberchondria severity

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be publicly shared due to privacy concerns and the sensitive nature of maternal and infant health information. However, anonymized data may be made available upon reasonable request to the corresponding author after publication of the study results.

REFERENCES:
- [Background] Boivin J, Takefman J, Braverman A. The fertility quality of life (FertiQoL) tool: development and general psychometric properties. Hum Reprod. 2011 Aug;26(8):2084-91. doi: 10.1093/humrep/der171. Epub 2011 Jun 10. PMID 21665875
- [Background] Brochu F, Robins S, Miner SA, Grunberg PH, Chan P, Lo K, Holzer HEG, Mahutte N, Ouhilal S, Tulandi T, Zelkowitz P. Searching the Internet for Infertility Information: A Survey of Patient Needs and Preferences. J Med Internet Res. 2019 Dec 12;21(12):e15132. doi: 10.2196/15132. PMID 31829963
- [Background] Buran, G., Toptaş Acar, B. The effect of social and emotional capacities on coping strategies and stress in infertile individuals. Curr Psychol 43, 29984-29994 (2024). https://doi.org/10.1007/s12144-024-06504-5
- [Background] Çakı, B., & Sohbet, R. (2021). The examination of reproductive information and stress levels of fertilite and infertile women. Adıyaman Üniversitesi Sağlık Bilimleri Dergisi, 7(1), 103-112.
- [Background] European Society of Human Reproduction and Embryology (ESHRE). (2021, August). Factsheet on infertility - prevalence, treatment and fertility decline in Europe.
- [Background] Irmak Vural P, Korpe G, Aslan E. Validity and Reliability of the Turkish Version of Screening Tool on Distress in Fertility Treatment (SCREENIVF). Psychiatr Danub. 2021 Dec;33(Suppl 13):278-287. PMID 35150496
- [Background] Mayette E, Scalise A, Li A, McGeorge N, James K, Mahalingaiah S. Assisted reproductive technology (ART) patient information-seeking behavior: a qualitative study. BMC Womens Health. 2024 Jun 15;24(1):346. doi: 10.1186/s12905-024-03183-z. PMID 38877503
- [Background] Verhaak CM, Lintsen AM, Evers AW, Braat DD. Who is at risk of emotional problems and how do you know? Screening of women going for IVF treatment. Hum Reprod. 2010 May;25(5):1234-40. doi: 10.1093/humrep/deq054. Epub 2010 Mar 13. PMID 20228392
- [Background] Starcevic V, Schimmenti A, Billieux J, Berle D. Cyberchondria in the time of the COVID-19 pandemic. Hum Behav Emerg Technol. 2021 Jan;3(1):53-62. doi: 10.1002/hbe2.233. Epub 2020 Nov 23. PMID 33363277